CLINICAL TRIAL: NCT03519776
Title: Variation of Progesterone in IVF Cycles
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 1710-MUS-106-LB
Record Dates: First submitted 2018-04-25; First posted 2018-05-09 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Progesterone Resistance
MeSH Terms: conditions — Progesterone Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn. Each blood sample will consist of 10 cc of blood, to be centrifuged and the serum shared into 3 vials before freezing at minus 20 degrees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Progesterone variation — The potential gain for medical caretakers and patients would be a certainty if the progesterone level is affected by variations during daytime

SUMMARY:
to examine if a natural daytime variation in progesterone levels may explain parts of the inconsistent findings from studies reporting divergent results concerning this matter and will be carried out by several blood samples from the same patient during the day of ovulation triggering.

DETAILED DESCRIPTION:
The impact of the progesterone level at the end of the follicular phase in stimulated IVF/ICSI cycles and its effect on the pregnancy rate and oocyte quality is controversial, which arises from conflicting results in retrospective studies and meta-analyses. This study is assumed to examine if a natural daytime variation in progesterone levels may explain parts of the inconsistent findings from studies reporting divergent results concerning this matter and will be carried out by several blood samples from the same patient during the day of ovulation triggering. If variation is present, the impact of variation on the developing oocyte and embryo quality will be estimated by embryo quality indicators.

ELIGIBILITY:
Inclusion Criteria:

* patients 18-45 years
* BMI 18-35 kg/m2
* Menstrual cycle length 24-35 days
* Stimulation with rFSH or hMG

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patient who will undergo IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
The variation of serum progesterone around the ovulation triggering in IVF-cycles | 6-8 months
  the circadian secretion-pattern of progesterone during early follicular phase of normal cycling females

CONTACTS AND LOCATIONS:
Overall Officials: Upma Shanker, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Venetis CA, Kolibianakis EM, Bosdou JK, Lainas GT, Sfontouris IA, Tarlatzis BC, Lainas TG. Estimating the net effect of progesterone elevation on the day of hCG on live birth rates after IVF: a cohort analysis of 3296 IVF cycles. Hum Reprod. 2015 Mar;30(3):684-91. doi: 10.1093/humrep/deu362. Epub 2015 Jan 12. PMID 25586787
- [Background] Venetis CA, Kolibianakis EM, Bosdou JK, Tarlatzis BC. Progesterone elevation and probability of pregnancy after IVF: a systematic review and meta-analysis of over 60 000 cycles. Hum Reprod Update. 2013 Sep-Oct;19(5):433-57. doi: 10.1093/humupd/dmt014. Epub 2013 Jul 4. PMID 23827986
- [Background] Griesinger G, Mannaerts B, Andersen CY, Witjes H, Kolibianakis EM, Gordon K. Progesterone elevation does not compromise pregnancy rates in high responders: a pooled analysis of in vitro fertilization patients treated with recombinant follicle-stimulating hormone/gonadotropin-releasing hormone antagonist in six trials. Fertil Steril. 2013 Dec;100(6):1622-8.e1-3. doi: 10.1016/j.fertnstert.2013.08.045. Epub 2013 Sep 29. PMID 24083873
- [Background] Requena A, Cruz M, Bosch E, Meseguer M, Garcia-Velasco JA. High progesterone levels in women with high ovarian response do not affect clinical outcomes: a retrospective cohort study. Reprod Biol Endocrinol. 2014 Jul 26;12:69. doi: 10.1186/1477-7827-12-69. PMID 25064138
- [Background] Yding Andersen C, Bungum L, Nyboe Andersen A, Humaidan P. Preovulatory progesterone concentration associates significantly to follicle number and LH concentration but not to pregnancy rate. Reprod Biomed Online. 2011 Aug;23(2):187-95. doi: 10.1016/j.rbmo.2011.04.003. Epub 2011 Apr 28. PMID 21665546
- [Background] Patton PE, Lim JY, Hickok LR, Kettel LM, Larson JM, Pau KY. Precision of progesterone measurements with the use of automated immunoassay analyzers and the impact on clinical decisions for in vitro fertilization. Fertil Steril. 2014 Jun;101(6):1629-36. doi: 10.1016/j.fertnstert.2014.02.037. Epub 2014 Mar 21. PMID 24661729
- [Background] Bungum L, Jacobsson AK, Rosen F, Becker C, Yding Andersen C, Guner N, Giwercman A. Circadian variation in concentration of anti-Mullerian hormone in regularly menstruating females: relation to age, gonadotrophin and sex steroid levels. Hum Reprod. 2011 Mar;26(3):678-84. doi: 10.1093/humrep/deq380. Epub 2011 Jan 11. PMID 21227943
- [Background] Bosch E, Labarta E, Crespo J, Simon C, Remohi J, Jenkins J, Pellicer A. Circulating progesterone levels and ongoing pregnancy rates in controlled ovarian stimulation cycles for in vitro fertilization: analysis of over 4000 cycles. Hum Reprod. 2010 Aug;25(8):2092-100. doi: 10.1093/humrep/deq125. Epub 2010 Jun 10. PMID 20539042
- [Background] Thomsen LH, Kesmodel US, Andersen CY, Humaidan P. Daytime Variation in Serum Progesterone During the Mid-Luteal Phase in Women Undergoing In Vitro Fertilization Treatment. Front Endocrinol (Lausanne). 2018 Mar 19;9:92. doi: 10.3389/fendo.2018.00092. eCollection 2018. PMID 29615975
- [Derived] Shanker U, Lawrenz B, Bungum L, Depret Bixio L, Ruiz F, Coughlan C, Fatemi HM. Significant Serum Progesterone Variations on the Day of Final Oocyte Maturation in Stimulated IVF Cycles. Front Endocrinol (Lausanne). 2019 Nov 20;10:806. doi: 10.3389/fendo.2019.00806. eCollection 2019. PMID 31824423